CLINICAL TRIAL: NCT07119281
Title: Effect of Retraction Techniques on Scan Accuracy
Brief Title: Gingival Retraction for Digital Scan Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Merve Benli, Assos.prof.dr.merve benli, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: mbenli; mbenli (Other: MUSC)
Record Dates: First submitted 2025-07-21; First posted 2025-08-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Data Accuracy, Bleeding Control
MeSH Terms: interventions — Astringents; Aluminum Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A: Cordless paste with astringent (EXP) (Experimental): gingival retraction model 1 Expasyl (Acteon PVT LTD)
  Interventions: Procedure: Group A: Cordless paste with astringent (EXP): Expasyl (Acteon PVT LTD)
- Group B: Cordless paste without astringent (MF): (Experimental): gingival retraction model 2 Magic FoamCord (Coltene Whaledent AG)
  Interventions: Procedure: Group B: Cordless paste without astringent (MF): Magic FoamCord (Coltene Whaledent AG)
- Group C:Laser troughing (LT): (Experimental): gingival retraction model 3 Diode laser (iLase; Biolase Inc.)
  Interventions: Procedure: Group C: Laser troughing (LT): Diode laser (iLase; Biolase Inc.)
- Retraction cord with astringent (RCA; Control group): (Other): control-Knitted cord impregnated with aluminum chloride (Ultrapak + Viscostat Clear; Ultradent Inc.)
  Interventions: Procedure: Group D: Retraction cord with astringent (RCA; Control group): Knitted cord impregnated with aluminum chloride (Ultrapak + Viscostat Clear; Ultradent Inc.)

INTERVENTIONS:
Procedure: Group A: Cordless paste with astringent (EXP): Expasyl (Acteon PVT LTD) — Chemical gingival retraction method
  Arms: Group A: Cordless paste with astringent (EXP)
Procedure: Group B: Cordless paste without astringent (MF): Magic FoamCord (Coltene Whaledent AG) — Chemical gingival retraction method
  Arms: Group B: Cordless paste without astringent (MF):
Procedure: Group C: Laser troughing (LT): Diode laser (iLase; Biolase Inc.) — Gingival retraction will be performed by using only laser. Cord will not be used.
  Arms: Group C:Laser troughing (LT):
Procedure: Group D: Retraction cord with astringent (RCA; Control group): Knitted cord impregnated with aluminum chloride (Ultrapak + Viscostat Clear; Ultradent Inc.) — Mechanical and chemical gingival retraction method will be used.
  Arms: Retraction cord with astringent (RCA; Control group):

SUMMARY:
The study aims to identify which retraction method offers optimal balance between tissue displacement, scan clarity, and patient comfort, particularly in the esthetic zone, while avoiding the use of CBCT. Results will guide clinicians in selecting the most effective and minimally invasive approach for digital impression workflows.

DETAILED DESCRIPTION:
This prospective clinical study investigates the impact of various gingival retraction techniques on scan accuracy, gingival displacement, bleeding control, and finish line visibility during intraoral scanning of anterior teeth. A total of 32 systemically and periodontally healthy participants were randomly assigned to one of five groups, each using a different retraction method:

1. Retraction cord with astringent (RCA; Control group): Knitted cord impregnated with aluminum chloride (Ultrapak + Viscostat Clear; Ultradent Inc.)
2. Cordless paste with astringent (EXP): Expasyl (Acteon PVT LTD)
3. Cordless paste without astringent (MF): Magic FoamCord (Coltene Whaledent AG)
4. Laser troughing (LT): Diode laser (iLase; Biolase Inc.)

Digital impressions were obtained before and after retraction using a Trios 3Shape intraoral scanner. The gingival displacement was measured digitally, and scan accuracy was analyzed via RMS error. Bleeding index, finish line visibility, and patient discomfort (VAS) were also recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age 25-40 years
2. Maxillary premolars with normal anatomical size, contour, and position
3. Systemically healthy individuals
4. Healthy gingiva and periodontium around abutments (GI = 0)
5. Good oral hygiene (PI = 0)
6. Pocket depth ≤ 3 mm
7. Thick gingival biotype

Exclusion Criteria:

1. Smokers
2. Systemic conditions affecting periodontal status
3. Attachment loss, bleeding on probing, or plaque accumulation

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2025-05-04 (Actual)

PRIMARY OUTCOMES:
gingival displacement | 30 days
  Vertical and horizontal gingival displacement before and after gingival retraction method will be measured by using digital caliper.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Medial University of South Carolina, Charleston, South Carolina
  - Medical University of South Carolina, College of Dental Medicine, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
patient's data obtained from study
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12/1/2025-21/1/2026